CLINICAL TRIAL: NCT01905592
Title: A Phase III, Randomized, Open Label, Multicenter, Controlled Trial of Niraparib Versus Physician's Choice in Previously-treated, HER2 Negative, Germline BRCA Mutation-positive Breast Cancer Patients
Brief Title: A Phase III Trial of Niraparib Versus Physician's Choice in HER2 Negative, Germline BRCA Mutation-positive Breast Cancer Patients
Acronym: BRAVO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to futility.
Sponsor: Tesaro, Inc. (Industry)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network); Breast International Group (Other); Myriad Genetic Laboratories, Inc. (Industry); US Oncology Research (Industry); Sarah Cannon (Industry); Facing Our Risk of Cancer Empowered (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 213551; 1307-BCG, BIG5-13 (Other: EORTC, BIG); PR-30-5010-C (Other: Tesaro)
Record Dates: First submitted 2013-07-18; First posted 2013-07-23 (Estimated); Results first posted 2020-08-27 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-10

CONDITIONS: Neoplasms, Breast; Carcinoma of Breast; Human Epidermal Growth Factor 2 Negative Carcinoma of Breast; BRCA1 Gene Mutation; BRCA2 Gene Mutation; Ovarian Neoplasms
Keywords: Human Epidermal Growth Factor 2 Negative Carcinoma of Breast; BRCA1 Gene Mutation; BRCA2 Gene Mutation; PARP Inhibitor; BRCA
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms | interventions — niraparib

STUDY DESIGN:
Intervention Model Description: Randomization will be 2:1 (treatment:control) in at least 215 patients with germline BRCA mutations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Physician's choice (Active Comparator): Physician may select from 4 active comparators
  Interventions: Drug: Physician's choice
- niraparib (Experimental): Patients will be randomized 2:1 to receive niraparib 300 mg (3x100 mg capsules) once daily for 21 continuous days
  Interventions: Drug: niraparib

INTERVENTIONS:
Drug: niraparib — 300 mg (3x100 mg capsules) once daily until progression or unacceptable toxicity develops
  Other Names: formerly MK-4827
  Arms: niraparib
Drug: Physician's choice — Choice of 4 standard of care metastatic breast cancer chemotherapies, until progression or unacceptable toxicity develops
  Arms: Physician's choice

SUMMARY:
The purpose of this study is to compare progression-free survival (PFS) in patients with advanced/metastatic breast cancer who have a BRCA mutation when treated with niraparib as compared to those treated with physician's choice

DETAILED DESCRIPTION:
This is a phase III, randomized, open label, multicenter, controlled trial of niraparib versus physician's choice in previously-treated, HER2 negative, germline BRCA mutation-positive breast cancer patients. Niraparib is an orally active PARP inhibitor. Niraparib (in a 2:1 ratio) will be administered once daily continuously during a 21-day cycle. Physician's choice will be administered on a 21-day cycle. Health-related quality of life will be measured. The safety and tolerability will be assessed by clinical review of adverse events (AEs), physical examinations, electrocardiograms (ECGs), and safety laboratory values.

ELIGIBILITY:
Inclusion Criteria:

1. Germline BRCA1 or BRCA2 mutation; patients with unknown BRCA status who meet NCCN BRCA screening criteria will be screened for BRCA mutation.
2. Histologically or cytologically confirmed HER2-negative metastatic or locally advanced disease that is not amenable to resection or radiation with curative intent.
3. Up to 2 prior cytotoxic regimens for advanced or metastatic breast cancer; patients with no prior cytotoxic regimens for advanced or metastatic disease will only be allowed if they relapsed during or within 12 months of (neo-) adjuvant cytotoxic therapy.
4. Prior therapy should have included a taxane and/or anthracycline (unless contraindication to those) in the neoadjuvant, adjuvant, or advanced/metastatic setting.

   a. Hormone receptor positive patients must also have hormone resistant disease; either relapsed while on adjuvant endocrine treatment, or within one year of completing adjuvant endocrine treatment, or progression on at least one line of endocrine treatment for advanced cancer.
5. ECOG performance status 0-2
6. Adequate bone marrow, kidney and liver function

Exclusion Criteria:

1. Patients with platinum resistant cancer
2. Symptomatic uncontrolled brain metastases
3. Prior diagnosis of Stage IV ovarian cancer; Stage III ovarian cancer must have a 5-year disease-free interval; Stage II ovarian cancer must have a 2-year disease-free interval
4. Known hypersensitivity to the components of niraparib
5. Invasive cancer other than breast cancer within 2 years (except basal or squamous cell carcinoma of the skin that has been definitely treated)
6. Pregnant or breast feeding patients
7. Immunocompromised patients
8. Known active Hepatitis B or C
9. Prior treatment with a PARP inhibitor
10. Known history of myelodysplastic syndrome (MDS).
11. known and persistent (>4 weeks) >/= grade 3 toxicity or fatigue from prior cancer treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2014-02-25 (Actual); Primary Completion 2018-05-23 (Actual); Study Completion 2021-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (98):
- United States (23):
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Clifton Park, New York
  - GSK Investigational Site, Lake Success, New York
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Webster, Texas
  - GSK Investigational Site, Weslaco, Texas
  - GSK Investigational Site, Low Moor, Virginia
  - GSK Investigational Site, Everett, Washington
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Green Bay, Wisconsin
- Belgium (5):
  - GSK Investigational Site, Aalst
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Liège
  - GSK Investigational Site, Namur
- Canada (4):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Kelowna, British Columbia
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- France (8):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Dijon
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Saint-Cloud
- Greece (5):
  - GSK Investigational Site, Heraklion,Crete
  - GSK Investigational Site, Marousi
  - GSK Investigational Site, Nea Kifissia
  - GSK Investigational Site, Neo Faliro
  - GSK Investigational Site, Thessaloniki
- Hungary (6):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Miskolc
  - GSK Investigational Site, Nyíregyháza
  - GSK Investigational Site, Pécs
  - GSK Investigational Site, Szeged
- GSK Investigational Site, Reykjavik, Iceland
- Israel (6):
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Holon
  - GSK Investigational Site, Kfar Saba
  - GSK Investigational Site, Rehovot
  - GSK Investigational Site, Tel Aviv
  - GSK Investigational Site, Tel Litwinsky
- Italy (11):
  - GSK Investigational Site, Lecce, Apulia
  - GSK Investigational Site, Meldola (FC), Emilia-Romagna
  - GSK Investigational Site, Parma, Emilia-Romagna
  - GSK Investigational Site, Rimini, Emilia-Romagna
  - GSK Investigational Site, Viterbo, Lazio
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Cremona, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Ancona, The Marches
  - GSK Investigational Site, Prato, Tuscany
  - GSK Investigational Site, Legnago (VR), Veneto
- Netherlands (3):
  - GSK Investigational Site, Leiden, RC
  - GSK Investigational Site, Limburg
  - GSK Investigational Site, Zwolle
- Poland (2):
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Racibórz
- Portugal (3):
  - GSK Investigational Site, Coimbra
  - GSK Investigational Site, Lisbon
  - GSK Investigational Site, Porto
- Spain (10):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Cáceres
  - GSK Investigational Site, L'Hospitalet de Llobregat
  - GSK Investigational Site, Lleida
  - GSK Investigational Site, Lugo
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Vigo
- United Kingdom (11):
  - GSK Investigational Site, Southampton, Hampshire
  - GSK Investigational Site, Northwood, Middlesex
  - GSK Investigational Site, Headington, Oxford, Oxfordshire
  - GSK Investigational Site, Sutton, Surrey
  - GSK Investigational Site, Bebington, Wirral
  - GSK Investigational Site, Belfast
  - GSK Investigational Site, Edinburgh
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, London
  - GSK Investigational Site, Nottingham
  - GSK Investigational Site, Whitchurch, Cardiff

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Facing our risk of cancer empowered website — http://www.facingourrisk.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Previously treated, human epidermal growth factor receptor 2 HER2 negative, germline Breast Cancer gene (gBRCA) mutation positive breast cancer participants were enrolled. The study was terminated due to futility.
Pre-assignment Details: Of the 216 participants enrolled, 1 participant was not randomized and 9 participants enrolled based on a local BRCA test results were later determined to be BRCA wild type by central testing. Therefore, only 206 of the 216 participants enrolled were included in the analysis, and were considered in centrally confirmed intent-to-treat (ITT) Population.
Groups:
- Physician's Choice: Physician selection from 4 standard of care metastatic breast cancer chemotherapies (eribulin or vinorelbine or gemcitabine or capecitabine), until progression or unacceptable toxicity develops.
- Niraparib: Niraparib 300 milligram (mg) (3x100 mg) capsules once daily until progression or unacceptable toxicity develops.
Period: Overall Study
Arm/Group | Physician's Choice | Niraparib
Started (Based on centrally confirmed intent-to-treat population) | 71 | 135
Completed (Based on centrally confirmed intent-to-treat population) | 0 | 0
Not Completed | 71 | 135
Not completed — Disease Progression | 51 | 110
Not completed — Toxicity | 1 | 16
Not completed — Physician Decision | 0 | 2
Not completed — Start of New anti-cancer Treatment | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Sponsor's decision | 1 | 1
Not completed — Not treated | 7 | 3
Not completed — Withdrawal by Subject | 10 | 2

BASELINE CHARACTERISTICS:
Population: The centrally-confirmed intent-to-treat population is defined as all randomized participants with a central confirmation of germline BRCA mutation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Physician's Choice | Niraparib | Total
Number analyzed (Participants) | 71 | 135 | 206
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 67 | 127 | 194
  65-74 years | 3 | 5 | 8
  >=75 years | 1 | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 135 | 203
  Male | 3 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 50 | 110 | 160
  Unknown or Not Reported | 15 | 19 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Ashkenazi Jewish descendant | 6 | 5 | 11
  Race: White or Caucasian | 59 | 108 | 167
  Race: Black | 3 | 6 | 9
  Race: Asian | 0 | 2 | 2
  Race: Unknown | 1 | 7 | 8
  Race: Missing | 2 | 7 | 9

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) - Central Review Assessment
Description: The primary objective of this study is to compare progression-free survival (PFS), as assessed by blinded central review, of participants with advanced/metastatic human epidermal growth factor receptor 2 (HER2)-negative gBRCA mutation breast cancer when treated with niraparib as compared to those treated with physician's choice single agent chemotherapy standards (eribulin, vinorelbine, gemcitabine or capecitabine). PFS is defined as the date of randomization to the date of disease progression or death due to any cause, whichever occurs earlier as per Response evaluation criteria in solid tumors (RECIST) version (v)1.1 as determined by central review assessment. Progressive Disease is defined as at least a 20 percent (%) increase in the sum of diameters of measured lesions taking as references the smallest sum of diameters recorded on study (including Baseline) and an absolute increase of >= 5 millimeter (mm).
Time Frame: From the date of randomization to the date of disease progression or death due to any cause, whichever occurs earlier, up to 4 years
Population: Centrally Confirmed intent-to-treat (ITT) Population is defined as all randomized participants with a central confirmation of germline BRCA mutation.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Physician's Choice | Niraparib
Number analyzed (Participants) | 71 | 135
Months | 3.1 [1.6 to 7.2] | 4.1 [2.9 to 4.5]

2. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) was defined as the time from randomization to the date of death of any causes.
Time Frame: From treatment randomization to date of death of any cause, up to 4 years
Population: Centrally Confirmed ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Physician's Choice | Niraparib
Number analyzed (Participants) | 71 | 135
Months | 15.8 [12.1 to 18.4] | 14.5 [11.7 to 17.2]

3. Secondary Outcome: Number of Participants With Central BRCA Mutation Status
Description: Blood samples were collected to evaluate central BRCA mutation status of participants. Baseline was defined as the most recent non-missing measurement prior to or on the first administration of study drug. Number of participants with central BRCA mutation status as BRCA1 positive only, BRCA2 positive only, Rearrangement only, BRCA1 and BRCA2 positive, BRCA1 positive and rearrangement, and BRCA2 positive and rearrangement were reported.
Time Frame: At Baseline (Cycle 1 Day1) (Cycle duration was 21 days)
Population: Centrally Confirmed ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Physician's Choice | Niraparib
Number analyzed (Participants) | 71 | 135
Participants
  BRCA1 positive only | 38 | 66
  BRCA2 positive only | 28 | 57
  Rearrangement only | 3 | 7
  BRCA1 and BRCA2 positive | 1 | 3
  BRCA1 positive and rearrangement | 1 | 1
  BRCA2 positive and rearrangement | 0 | 1

4. Secondary Outcome: Number of Participants With Serious Adverse Events (SAE) and Non-serious Adverse Events (Non-SAE)
Description: An adverse event (AE) is any untoward medical occurrence that occurs in a participant or clinical investigation participant administered a pharmaceutical product, and which does not necessarily have to have a causal relationship with this treatment. An SAE is defined as any untoward medical occurrence or effect in a participant, whether or not considered related to the protocol treatment, at any dose that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing participant hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, is an medically important event or reaction as per medical and scientific judgment. Adverse events which were not serious adverse events were considered as non serious adverse events.
Time Frame: Up to 7 years
Population: Safety Population comprised of all participants who started their allocated treatment (received at least one dose of allocated drug). Only those participants with data available at specified time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Physician's Choice | Niraparib
Number analyzed (Participants) | 65 | 134
Participants
  SAE | 4 | 33
  Non-SAE | 62 | 134

5. Secondary Outcome: Progression Free Survival (PFS) - Investigator Assessment
Description: PFS is defined as the date of randomization to the date of disease progression or death due to any cause, whichever occurs earlier as per RECIST version 1.1 as determined by Investigator assessment. Progressive Disease is defined as at least a 20 % increase in the sum of diameters of measured lesions taking as references the smallest sum of diameters recorded on study (including Baseline) and an absolute increase of >= 5 mm.
Time Frame: Assessed up to 4 years
Population: Centrally confirmed ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Physician's Choice | Niraparib
Number analyzed (Participants) | 71 | 135
Months | 3.1 [2.7 to 5.1] | 5.0 [4.2 to 5.5]

6. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure was defined from the date of randomization to progression or discontinuation of treatment for any reason, including but not restricted to disease progression, treatment toxicity and death.
Time Frame: Date of randomization to discontinuation of treatment for any reason, up to 4 years
Population: Centrally Confirmed ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Physician's Choice | Niraparib
Number analyzed (Participants) | 71 | 135
Months | 2.6 [1.6 to 3.2] | 4.3 [4.0 to 5.5]

7. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of the participants who achieved a complete response (CR) or partial response (PR) to treatment evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Complete Response (CR)=disappearance of all target and non-target lesions and normalization of tumor markers. Pathological lymph nodes must have short axis measures <10 mm. Partial Response (PR)= at least a 30% decrease in the sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of target lesions, taking as reference the Baseline sum of diameters. Percentage values are rounded off up to 1 decimal.
Time Frame: Up to 4 years
Population: Centrally Confirmed ITT population. Only those participants with confirmed response were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Physician's Choice | Niraparib
Number analyzed (Participants) | 64 | 126
Percentage of participants | 12.5 [5.6 to 23.2] | 21.4 [14.6 to 29.6]

8. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response was defined as the time from first documentation of response (confirmed CR or PR) until the time of first documentation of disease progression by RECIST v1.1 or death by any cause.
Time Frame: Up to 4 years
Population: Centrally Confirmed ITT population. Only those participants with confirmed response were analyzed.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Physician's Choice | Niraparib
Number analyzed (Participants) | 64 | 126
Months | 5.65 [5.65 to 14.78] | 4.14 [2.79 to 6.90]

9. Other Pre Specified Outcome: Number of Participants With Minimally Clinically Important Difference (MCID) Status in European Organization for Research and Treatment of Cancer-Quality of Life Questionnaire-C30 (EORTC-QLQ-C30)
Description: The number of participants with MCID status in EORTC-QLQ-C30 was planned to be evaluated.The EORTC- QLQ-C30 includes 30-items with single and multi-item scales. These include five functional scales (physical functioning, role functioning cognitive functioning, emotional functioning and social functioning), three symptom scales (fatigue, pain and nausea/vomiting), a global health status (GHS)/ Quality-of-Life (QoL) scale, and six single items (constipation, diarrhea, insomnia, dyspnea, appetite loss and financial difficulties). Response options are 1 to 4. The average score can be transformed to 0 to 100, a high score for functional scales/ GHS/QoL represents better functioning ability or health-related quality-of-life (HRQoL), whereas a high score for symptom scales/ single items represents significant symptomatology.
Time Frame: Up to 7 years
Population: ITT Population comprised of all randomized participants. This was an other pre-specified outcome measure. The results for this outcome measure will never be posted.
Arm/Group | Physician's Choice | Niraparib
Number analyzed (Participants) | 0 | 0

10. Other Pre Specified Outcome: Number of Participants With Euroqol 5 Dimension 5 Level (EQ-5D-5L) Dimension Scores by Visit
Description: The number of participants with EQ-5D-5L scores by visit were planned to be evaluated. EQ-5D-5L is self-assessment questionnaire, consisting of 5 items covering 5 dimensions (mobility,self care, usual activities, pain/discomfort and anxiety/depression). Each dimension is measured by 5-point Likert scale(no problems, slight problems, moderate problems, severe problems and extreme problems). Responses for 5 dimensions together formed a 5-figure description of health state (e.g.11111 indicates no problems in all 5 dimensions). Each of these 5 figure health states were to be converted to a single index score. Range for EQ-5D-5L index score is 0 (worst health) to 100 (best health), higher the score better the health status.
Time Frame: Up to 7 years
Population: ITT Population. This was an other pre-specified outcome measure. The results for this outcome measure will never be posted.
Arm/Group | Physician's Choice | Niraparib
Number analyzed (Participants) | 0 | 0

11. Other Pre Specified Outcome: Number of Participants With Any Subsequent Therapies Post Discontinuation of Study Treatment and Association With Potential Survival Related Outcomes
Description: The number of participants with any subsequent therapies post-discontinuation of study treatment and association with potential survival related outcomes were planned to be evaluated.
Time Frame: Up to 7 years
Population: Safety Population. This was an other pre-specified outcome measure. The results for this outcome measure will never be posted.
Arm/Group | Physician's Choice | Niraparib
Number analyzed (Participants) | 0 | 0

12. Other Pre Specified Outcome: Number of Participants With Presence of Genetic and Non-genetic Biomarkers
Description: Biomarkers include germline and tumor mutations including somatic BRCA1 and 2 mutations, reversion mutations, loss of heterozygosity as well as genome landscape and transcriptional or functional measures of homologous recombination (HR) deficiency were planned to be evaluated.
Time Frame: Up to 7 years
Population: Centrally Confirmed ITT Population. This was an other pre-specified outcome measure. The results for this outcome measure will never be posted.
Arm/Group | Physician's Choice | Niraparib
Number analyzed (Participants) | 0 | 0

13. Other Pre Specified Outcome: Number of Participants With Germline BRCA1 and BRCA2 Mutation Status in Association With Survival Related Outcomes
Description: Participants with germline BRCA1 and BRCA2 mutation status in association with survival related outcomes were planned to be evaluated.
Time Frame: Up to 7 years
Population: as for outcome 12
Arm/Group | Physician's Choice | Niraparib
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Number of Participants With Serious Adverse Events Related to New Malignancy
Description: The number of participants with serious adverse events related to new malignancy were reported.
Time Frame: Up to 7 years
Population: Safety Population. Only those participants with data available at specified time were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Physician's Choice | Niraparib
Number analyzed (Participants) | 65 | 134
Participants | 0 | 2

15. Secondary Outcome: Number of Participants With Subsequent Anticancer Therapies
Description: The number of participants with subsequent anticancer therapies were evaluated. Data has been reported as per following categories: any new anitumoral therapy, any chemotherapy, any radiotherapy, any surgery, any hormonal therapy, any targeted agents, and any other treatment. Participants may have received more than one subsequent therapies.
Time Frame: Up to 7 years
Population: Safety Population. Only those participants with data available at specified time were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Physician's Choice | Niraparib
Number analyzed (Participants) | 65 | 134
Participants
  Any new antitumoral therapy | 55 | 108
  Any chemotherapy | 48 | 96
  Any radiotherapy | 22 | 48
  Any surgery | 5 | 13
  Any hormonal therapy | 13 | 27
  Any targeted agent therapy | 19 | 22
  Any other treatment | 8 | 17

ADVERSE EVENTS:
Time Frame: All-cause mortality, Serious adverse events (SAEs) and non-serious AEs (non-SAEs) were collected up to 7 years
Description: Safety Population was used to assess SAEs and non-SAEs, which comprised of all participants who started their allocated treatment (received at least one dose of allocated drug). Seven participants from Centrally Confirmed (ITT) Population (N=206) did not receive study treatment, hence was not included in Safety Population (N=199).
Arm/Group | Physician's Choice | Niraparib
All-Cause Mortality (participants affected / at risk) | 39/65 | 79/134
Serious Adverse Events (participants affected / at risk) | 4/65 | 33/134
Other Adverse Events (participants affected / at risk) | 62/65 | 134/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physician's Choice (N=65) | Niraparib (N=134)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 10 (29)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 9 (19)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 5 (5)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 4 (5)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (2) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Language disorder (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Platelet count decreased (Investigations) | 0 (0) | 2 (3)
Electrocardiogram ST segment depression (Investigations) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (2)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physician's Choice (N=65) | Niraparib (N=134)
Anaemia (Blood and lymphatic system disorders) | 23 (63) | 91 (396)
Nausea (Gastrointestinal disorders) | 24 (36) | 82 (141)
Fatigue (General disorders) | 29 (49) | 66 (121)
Weight decreased (Investigations) | 10 (12) | 53 (97)
Vomiting (Gastrointestinal disorders) | 11 (16) | 51 (77)
Constipation (Gastrointestinal disorders) | 11 (13) | 48 (74)
Headache (Nervous system disorders) | 10 (11) | 44 (75)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (9) | 48 (155)
Decreased appetite (Metabolism and nutrition disorders) | 7 (10) | 41 (56)
Platelet count decreased (Investigations) | 3 (5) | 43 (90)
Neutropenia (Blood and lymphatic system disorders) | 19 (43) | 27 (64)
Diarrhoea (Gastrointestinal disorders) | 22 (30) | 19 (24)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (9) | 29 (42)
Neutrophil count decreased (Investigations) | 10 (15) | 26 (66)
White blood cell count decreased (Investigations) | 5 (12) | 32 (83)
Asthenia (General disorders) | 9 (11) | 24 (61)
Dizziness (Nervous system disorders) | 6 (9) | 26 (35)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (12) | 25 (35)
Insomnia (Psychiatric disorders) | 4 (5) | 25 (32)
Anxiety (Psychiatric disorders) | 8 (9) | 18 (24)
Abdominal pain (Gastrointestinal disorders) | 10 (12) | 14 (21)
Alanine aminotransferase increased (Investigations) | 7 (10) | 18 (26)
Gamma-glutamyltransferase increased (Investigations) | 7 (16) | 17 (28)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (6) | 19 (24)
Abdominal pain upper (Gastrointestinal disorders) | 3 (5) | 17 (24)
Blood alkaline phosphatase increased (Investigations) | 5 (8) | 15 (25)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 15 (17)
Leukopenia (Blood and lymphatic system disorders) | 9 (40) | 11 (35)
Stomatitis (Gastrointestinal disorders) | 6 (7) | 14 (20)
Pyrexia (General disorders) | 4 (8) | 16 (25)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 13 (17)
Hypertension (Vascular disorders) | 1 (1) | 17 (38)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (10) | 16 (34)
Oedema peripheral (General disorders) | 6 (9) | 9 (10)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (7) | 9 (11)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 12 (31) | 0 (0)
Lymphocyte count decreased (Investigations) | 4 (6) | 9 (31)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 10 (12)
Tachycardia (Cardiac disorders) | 2 (3) | 11 (11)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 9 (9)
Weight increased (Investigations) | 7 (7) | 6 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 10 (10)
Dry mouth (Gastrointestinal disorders) | 5 (5) | 6 (7)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 7 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5)
Paraesthesia (Nervous system disorders) | 6 (6) | 5 (5)
Urinary tract infection (Infections and infestations) | 3 (3) | 7 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (8) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 9 (10)
Influenza like illness (General disorders) | 2 (5) | 8 (9)
Pain (General disorders) | 1 (1) | 7 (7)
Ill-defined disorder (General disorders) | 4 (11) | 6 (8)
Mucosal inflammation (General disorders) | 4 (4) | 2 (2)
Blood creatinine increased (Investigations) | 4 (5) | 6 (7)
Lethargy (Nervous system disorders) | 4 (7) | 5 (5)
Hypoaesthesia (Nervous system disorders) | 5 (5) | 4 (7)
Depression (Psychiatric disorders) | 0 (0) | 7 (7)
Hot flush (Vascular disorders) | 0 (0) | 7 (8)
Lymphoedema (Vascular disorders) | 4 (11) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 9 (9)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (8)
Erythema (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (4)
Nasopharyngitis (Infections and infestations) | 3 (3) | 8 (12)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 8 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 7 (11)

LIMITATIONS AND CAVEATS:
IDMC interim analysis concluded that concerns with the quantity and quality of data in the control arm precluded meaningful comparative analyses and generation of a clinically useful endpoint, therefore enrollment was ended prematurely.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-01-20): https://cdn.clinicaltrials.gov/large-docs/92/NCT01905592/Prot_002.pdf
  • Statistical Analysis Plan (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/92/NCT01905592/SAP_003.pdf